CLINICAL TRIAL: NCT02318212
Title: International Observational E-Registry on the Use of Dilapan-S/Dilasoft Osmotic Dilators for Cervical Priming Prior to Induced Abortion
Brief Title: Dilapan-S / Dilasoft E-Registry in Induced Abortion
Acronym: DSREGISTRYIA
Status: Completed | Type: Observational
Sponsor: Medicem International CR s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIS-2014-010
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Abortion, Induced
Keywords: Cervical dilatation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dilapan-S — Synthetic osmotic dilators Dilapan-S or Dilasoft for cervical priming prior to induced abortion
  Other Names: Dilasoft

SUMMARY:
International Observational E-Registry on the use of osmotic dilators DILAPAN-S® / DILASOFT® for cervical priming prior to induced abortion.

DETAILED DESCRIPTION:
International, multicentre, non-interventional, observational e-registry, post market clinical follow up study to document current clinical use of Dilapan-S or Dilasoft for cervical priming before induced abortion with regard to the number of dilators used, duration of insertion of dilators in situ and unusual complications consequent of their use.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy ≥ 6 and ≤ 24 weeks gestation
* Patients who are capable of giving consent and sign the form
* Abortion being made in compliance with the Abortion Act 1967 (For England, Wales and Scotland)

Exclusion Criteria:

* Clinical signs of uterine, vaginal or vulvar infection
* Acute bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients indicated for cervical priming with Dilapan-S or Dilasoft prior to induced abortion and meet all inclusion and exclusion criteria in centres involved in data collection.
Sampling Method: Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of inserted osmotic dilators | max. up to 24 hrs; estimated average 6 hrs
Total time taken for cervical priming with Dilapan-S/Dilasoft | max. up to 24 hrs; estimated average 6 hrs
  Duration of leaving osmotic dilators in situ

SECONDARY OUTCOMES:
Type of synthetic osmotic dilator used | max. up to 24 hrs; estimated average 6 hrs
  Dilapan-S or Dilasoft
Complications during cervical priming | up to 24 hrs; estimated average 6 hrs
  pre-operative bleeding, fever, pain, nausea, vomiting, diarrhoea, premature passage of foetal or chorionic tissue
Other observed undesirable effects uf use of synthetic osmotic dilators | up to 24 hrs; estimated average 6 hrs
Need of additional mechanical dilation | up to 10 minutes after osmotic dilators extraction
  In cases, when surgical abortion is performed
Surgical operative time | estimated max. up to 10 min, estimated average 8 min.
  Period from speculum insertion in to speculum extraction out
Initiation-to-delivery time | hrs
  In case of medical abortion
Induction-to-delivery time | up to 72 hrs; estimated average 48 hrs
  In case of medical abortion
Complications related to induced abortion procedure | up to 24 hrs; estimated average 12 hrs
Infectious complication and its relation to the use of Dilapan-S/Dilasoft | up to 72 hrs; Complications, if any, will be followed-up until stable situation has been reached.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lohr, MD, Principal Investigator — British Pregnancy Advisory Service, UK; Jiri Hanacek, MD, Principal Investigator — Institute of Care for Mother and Child, Prague, CZ; Natalia Kan, Prof., MD, Principal Investigator — Research Center for Obstetrics, Gynecology and Perinatology, Moscow; John Roizin, MD, Principal Investigator — Allentown Women´s Center, Bethlehem, PA, US; Mary Jane Bovo, MD, Principal Investigator — Choices Women´s Medical Center, New York; LeRoy Carhart, MD, Principal Investigator — Germantown Reproductive Health Service

REFERENCES:
- [Background] Allen RH, Goldberg AB; Board of Society of Family Planning. Cervical dilation before first-trimester surgical abortion (<14 weeks' gestation). SFP Guideline 20071. Contraception. 2007 Aug;76(2):139-56. doi: 10.1016/j.contraception.2007.05.001. Epub 2007 Jul 10. PMID 17656184
- [Background] Fox MC, Krajewski CM. Cervical preparation for second-trimester surgical abortion prior to 20 weeks' gestation: SFP Guideline #2013-4. Contraception. 2014 Feb;89(2):75-84. doi: 10.1016/j.contraception.2013.11.001. Epub 2013 Nov 11. PMID 24331860
- [Background] Newmann S, Dalve-Endres A, Drey EA; Society of Family Planning. Clinical guidelines. Cervical preparation for surgical abortion from 20 to 24 weeks' gestation. Contraception. 2008 Apr;77(4):308-14. doi: 10.1016/j.contraception.2008.01.004. Epub 2008 Mar 4. PMID 18342657
- [Background] Schulz KF, Grimes DA, Cates W Jr. Measures to prevent cervical injury during suction curettage abortion. Lancet. 1983 May 28;1(8335):1182-5. doi: 10.1016/s0140-6736(83)92464-9. PMID 6133988
- [Background] Lichtenberg ES. Complications of osmotic dilators. Obstet Gynecol Surv. 2004 Jul;59(7):528-36. doi: 10.1097/00006254-200407000-00022. PMID 15199271
- [Background] Samuel MI, Parsons JH. Hygroscopic dilator (Dilapan-S) and misoprostol combination for the early first-trimester termination of pregnancy: a pilot study. J Fam Plann Reprod Health Care. 2009 Jan;35(1):45-7. doi: 10.1783/147118909787072234. PMID 19126319
- [Background] Chambers DG, Willcourt RJ, Laver AR, Baird JK, Herbert WY. Comparison of Dilapan-S and laminaria for cervical priming before surgical pregnancy termination at 17-22 weeks' gestation. Int J Womens Health. 2011;3:347-52. doi: 10.2147/IJWH.S25551. Epub 2011 Oct 20. PMID 22114527
- [Background] Chen FC, Bergann A, Krosse J, Merholz A, David M. Isosorbide mononitrate vaginal gel versus misoprostol vaginal gel versus Dilapan-S for cervical ripening before first trimester curettage. Eur J Obstet Gynecol Reprod Biol. 2008 Jun;138(2):176-9. doi: 10.1016/j.ejogrb.2007.09.009. Epub 2007 Nov 5. PMID 17980952
- [Background] Bartz D, Maurer R, Allen RH, Fortin J, Kuang B, Goldberg AB. Buccal misoprostol compared with synthetic osmotic cervical dilator before surgical abortion: a randomized controlled trial. Obstet Gynecol. 2013 Jul;122(1):57-63. doi: 10.1097/AOG.0b013e3182983889. PMID 23743471
- [Background] Lyus R, Lohr PA, Taylor J, Morroni C. Outcomes with same-day cervical preparation with Dilapan-S osmotic dilators and vaginal misoprostol before dilatation and evacuation at 18 to 21+6 weeks' gestation. Contraception. 2013 Jan;87(1):71-5. doi: 10.1016/j.contraception.2012.07.006. Epub 2012 Aug 13. PMID 22898362
- [Background] Poon LC, Parsons J. Audit of the effectiveness of cervical preparation with Dilapan prior to late second-trimester (20-24 weeks) surgical termination of pregnancy. BJOG. 2007 Apr;114(4):485-8. doi: 10.1111/j.1471-0528.2006.01257.x. Epub 2007 Feb 19. PMID 17309543
- [Background] Newmann SJ, Sokoloff A, Tharyil M, Illangasekare T, Steinauer JE, Drey EA. Same-day synthetic osmotic dilators compared with overnight laminaria before abortion at 14-18 weeks of gestation: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):271-278. doi: 10.1097/AOG.0000000000000080. PMID 24402587